CLINICAL TRIAL: NCT00803829
Title: Synbiotic Treatment of Ulcerative Colitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: National Association for Colitis and Crohn's Disease (Other)
Responsible Party: Professor George Macfarlane, University of Dundee
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 20509; NACC: M/08/2; REC: 08/S1402/45; RD: 2007GA08
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-07

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Synbiotics; Prebiotics; Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Synbiotic (Synergy1/B. longum) — Probiotic Bifidobacterium longum Prebiotic Synergy 1
  Other Names: prebiotic; probiotic

SUMMARY:
Ulcerative colitis (UC) is one of the two main forms of inflammatory bowel disease. UC is associated with high morbidity and incurs significant social, commercial and NHS costs. For a variety of reasons, many patients are refractile to standard therapies, which often have undesirable side-effects. However, an inexpensive and non-toxic treatment based on the synbiotic concept may prove to be effective in these individuals. A synbiotic is a mixture of a probiotic (a live microorganism) and a prebiotic, which is a carbohydrate that serves as a food source for the probiotic, allowing it to grow better in the gut. The aim of this study is to determine whether a synbiotic comprised of fructooligosaccharides and inulin, together with a bifidobacterial probiotic (Bifidobacterium longum), that we have previously shown to reduce inflammatory processes in the gut wall (mucosa) in a short-term pilot trial, can colonise the bowel, reduce mucosal inflammation, and induce remission in UC patients with active disease. It is planned to establish a double-blinded, controlled, randomised investigation involving 46 patients for six months. If the results from our pilot study can be reproduced and maintained in a long-term investigation, the synbiotic could become available very quickly, and would provide an inexpensive and effective treatment for UC, making a significant contribution to relieving the clinical and financial burdens of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative colitis
* Stable doses of medications for UC for the preceding three months
* Mayo score of 6 to 12
* Sigmoidoscopy subscore of 2
* Stable doses of medication

Exclusion Criteria:

* Pregnancy
* Lactation
* Antibiotic therapy in the last three months
* Probiotic or prebiotic therapy in the last month
* Crohn's Disease, indeterminate colitis
* Alterations to medications in the last three months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Reduction in mucosal TNF-alpha | 6 months

SECONDARY OUTCOMES:
Induction of clinical remission measured by a reduction in Mayo disease activity score | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: George Macfarlane, PhD, Principal Investigator — University of Dundee; Sandra Macfarlane, PhD, Principal Investigator — University of Dundee; Nigel Reynolds, BA(Hons) MBChB FRCP, Principal Investigator — Tayside University Hospitals Trust; Craig Mowatt, Principal Investigator — Tayside University Hospital Trust; John Dillon, Principal Investigator — University of Dundee
Locations (1):
- Ninewells Hospital and Medical School, Dundee, Tayside, United Kingdom

REFERENCES:
- [Background] Macfarlane S, Furrie E, Cummings JH, Macfarlane GT. Chemotaxonomic analysis of bacterial populations colonizing the rectal mucosa in patients with ulcerative colitis. Clin Infect Dis. 2004 Jun 15;38(12):1690-9. doi: 10.1086/420823. Epub 2004 May 25. PMID 15227614
- [Background] Furrie E, Macfarlane S, Kennedy A, Cummings JH, Walsh SV, O'neil DA, Macfarlane GT. Synbiotic therapy (Bifidobacterium longum/Synergy 1) initiates resolution of inflammation in patients with active ulcerative colitis: a randomised controlled pilot trial. Gut. 2005 Feb;54(2):242-9. doi: 10.1136/gut.2004.044834. PMID 15647189
- [Background] Fite A, Macfarlane GT, Cummings JH, Hopkins MJ, Kong SC, Furrie E, Macfarlane S. Identification and quantitation of mucosal and faecal desulfovibrios using real time polymerase chain reaction. Gut. 2004 Apr;53(4):523-9. doi: 10.1136/gut.2003.031245. PMID 15016746
- [Background] Furrie E, Macfarlane S, Cummings JH, Macfarlane GT. Systemic antibodies towards mucosal bacteria in ulcerative colitis and Crohn's disease differentially activate the innate immune response. Gut. 2004 Jan;53(1):91-8. doi: 10.1136/gut.53.1.91. PMID 14684582
- [Background] Steed H, Macfarlane GT, Macfarlane S. Prebiotics, synbiotics and inflammatory bowel disease. Mol Nutr Food Res. 2008 Aug;52(8):898-905. doi: 10.1002/mnfr.200700139. PMID 18383235
- [Background] Macfarlane GT, Steed H, Macfarlane S. Bacterial metabolism and health-related effects of galacto-oligosaccharides and other prebiotics. J Appl Microbiol. 2008 Feb;104(2):305-44. doi: 10.1111/j.1365-2672.2007.03520.x. PMID 18215222